CLINICAL TRIAL: NCT07028281
Title: A Multicenter, Open-label, Phase II Clinical Study of SHR-4849 Injection Combined With Other Antineoplastic Drugs in Patients With Malignant Solid Tumors
Brief Title: A Trial of SHR-4849 Combined With Other Antitumor Drugs in Patients With Malignant Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4849-201
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-4849、SHR-1316、SHR-8068、BP102、carboplatin、cisplatin

INTERVENTIONS:
Drug: SHR-4849、SHR-1316、SHR-8068、BP102、carboplatin、cisplatin — SHR-4849、SHR-1316、SHR-8068、BP102、carboplatin、cisplatin

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-4849 injection combined with other antitumor drugs in patients with malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent prior to initiation of any study-procedures
2. Age from 18 to 75 years old at the time of signing the informed consent
3. Histologically or cytologically confirmed solid tumors
4. At least one measurable lesion was identified per RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Has a life expectancy of at least 3 months.
7. Adequate organ function
8. Subjects of both genders of child-bearing potential were required to use highly effective contraception from the time they provided written informed consent until 8 months after the last dose of the trial drug

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) metastasis.
2. Subjects with a history of malignant tumors within 5 years prior to the first dose
3. Subjects with uncontrolled cancer pain.
4. Subjects with severe cardiovascular disease.
5. Subjects with clinically significant hemorrhage
6. Subjects with uncontrolled pleural effusion, peritoneal effusion and pericardial effusion
7. Subjects highly suspected of interstitial lung disease
8. Subjects with serious infection within 4 weeks prior to the first dose
9. Known history of human immunodeficiency virus (HIV)，active hepatitis B virus or hepatitis C virus infection.
10. The adverse events of previous antineoplastic therapy did not recover to NCI-CTCAE≤ grade 1
11. Subjects who received anti-cancer treatment within 4 weeks prior to the first dose
12. Subjects who received major surgery within 4 weeks prior to the first dose
13. Subjects who plan to receive or have received live vaccines within 28 days prior to the first dose.
14. Female subjects who were pregnant, lactating, or planned to become pregnant during the study period
15. Known allergic to any component of investigational drugs
16. Alcohol abuse, drug abuse, other serious medical conditions (including mental illness) requiring combined treatment, and other conditions that may affect subject safety or data collection.
17. Based on the investigator's judgment, subjects with other conditions that may affect study results, interfere with study procedures,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
DLT：the incidence of events associated with the investigational drug determined by the investigator during the observation period(The first stage) | up to 21 days
Incidence and severity of AE/SAE：According to NCI-CTCAE v5.0 evaluation criteria, from the signing of informed consent to the end of safety follow-up(The first stage) | up to 24 months
Objective Response Rate (ORR) as Assessed by investigators(The second stage) | up to 24 months

SECONDARY OUTCOMES:
ORR(The first stage) | up to 24 months
  Objective Response Rate (ORR) as Assessed by investigators. The proportion of subjects whose best response was PR or CR according to RECIST1.1
DoR(The first stage) | up to 24 months
  Duration of Response (DOR) as Assessed by investigators according to RECIST1.1, Defined as the period of time from the first documented tumor response to the first documented objective progression or death of any cause.
DCR(The first stage) | up to 24 months
  Disease Control Rate(DCR) as Assessed by investigators. the proportion of subjects whose best response was PR or CR or SD according to RECIST1.1
PFS(The first stage) | up to 24 months
  Progression-free Survival (PFS) as Assessed by investigators according to RECIST1.1. Defined as the time from the initiation of the first medication to tumor progression or death from any cause (whichever comes first)
OS(The first stage) | up to 30 months
  Overall Survival . Defined as the time from the initiation of the first medication to death from any cause.
DoR(The second stage) | up to 24 months
  Duration of Response (DOR) as Assessed by investigators according to RECIST1.1, Defined as the period of time from the first documented tumor response to the first documented objective progression or death of any cause.
DCR(The second stage) | up to 24 months
  Disease Control Rate(DCR) as Assessed by investigators. the proportion of subjects whose best response was PR or CR or SD according to RECIST1.1
PFS(The second stage) | up to 24 months
  Progression-free Survival (PFS) as Assessed by investigators according to RECIST1.1. Defined as the time from the initiation of the first medication to tumor progression or death from any cause (whichever comes first)
OS(The second stage) | up to 30 months
  Overall Survival . Defined as the time from the initiation of the first medication to death from any cause.
Incidence and severity of AE/SAE：According to NCI-CTCAE v5.0 evaluation criteria, from the signing of informed consent to the end of safety follow-up(The second stage) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided